CLINICAL TRIAL: NCT01833650
Title: A Randomized Controlled Trial of the Effectiveness of Candy and Honey in Decreasing Salivary Gland Damage Following Radioiodine Therapy for Thyroid Cancer
Brief Title: The Use of Candy and Honey in Decreasing Salivary Gland Damage Following Radioiodine Therapy for Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: Bank of Cyprus Oncology Centre (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Assistant Professor of Oncology and Palliative Care, Cyprus University of Technology
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: AC-HCS-89
Record Dates: First submitted 2013-04-11; First posted 2013-04-17 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; radioiodine treatment; xerostomia; sialadenitis
MeSH Terms: conditions — Thyroid Neoplasms; Xerostomia; Sialadenitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard care (No Intervention): This arm represents the current standard care in patients with thyroid cancer undergoing radioiodine.
- Candy plus thymus honey mouthwash 12 (Experimental): This arm will consist 30 patients and will be the one of the intervention groups where each patient will be instructed to suck 1 or 2 lemon candies every 2-3 h in the daytime plus 4 thymus honey mouthwashes in between (at least one hour after the candy sucking) starting 12 hours after the ingestion of 131I therapy and for a duration of no more than 4 days.
  Interventions: Dietary Supplement: thymus honey mouthwash
- Candy plus thymus honey mouthwash 24 (Experimental): This arm will consist 30 patients and will be the one of the intervention groups where each patient will be instructed to suck 1 or 2 lemon candies every 2-3 h in the daytime plus 4 thymus honey mouthwashes in between (at least one hour after the candy sucking) starting 24 hours after the ingestion of 131I therapy and for a duration of no more than 4 days.
  Interventions: Dietary Supplement: thymus honey mouthwash
- Candy plus thymus honey mouthwash 1 (Experimental): This arm will consist 30 patients and will be the one of the intervention groups where each patient will be instructed to suck 1 or 2 lemon candies every 2-3 h in the daytime plus 4 thymus honey mouthwashes in between (at least one hour after the candy sucking) starting immediate after the ingestion of 131I therapy (about 1 hour) and for a duration of no more than 4 days
  Interventions: Dietary Supplement: thymus honey mouthwash

INTERVENTIONS:
Dietary Supplement: thymus honey mouthwash
  Arms: Candy plus thymus honey mouthwash 1; Candy plus thymus honey mouthwash 12; Candy plus thymus honey mouthwash 24

SUMMARY:
The purpose of this study is to determine whether the use of honey mouthwashes in the prevention of salivary side effects of 131I (radioiodine) therapy.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* They had a histological diagnosis of papillary, follicular, medullary or anaplastic thyroid cancer
* They had undergone total thyroidectomy
* They were able to provide consent

Exclusion Criteria:

* patients who had distant metastases,
* a history of salivary-gland disorders,
* collagen tissue disease
* diabetes mellitus,
* previous radioiodine therapy or external radiation to the head or neck
* allergy to the honey

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Grade of sialadenitis | Change from Baseline grade of sialadenitis at 6 and 24 months

SECONDARY OUTCOMES:
Grade of Xerostomia | Change from Baseline grade of xerostomia at 6 and 24 months
Level of Health related quality of life | Change from Baseline level of health related quality of life at 6 and 24 months

OTHER OUTCOMES:
Salivary Quantity (Quantitative Salivary Scintigraphy) | Change from Baseline quantity of saliva at 6 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Charalambous, PhD, Principal Investigator — Cyprus University of Technology
Locations (1):
- Bank of Cyprus Oncology, Nicosia, Cyprus